CLINICAL TRIAL: NCT05869032
Title: Establishing Normative Values for Event Related Potentials (ERPs) and Quantitative EEG (QEEG) in Adult, Healthy Volunteers
Brief Title: Normative QEEG/ERP Data for Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: Neuronetrix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SRP-1951
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Brain Function; Normative Values; Event-Related Potentials (ERP); Quantitative Electroencephalography (QEEG); Cognitive Processing; Frequency; Amplitude; Brain Activity; Electroencephalogram; Neural Processing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- Cohort 1 (n=10): Gender: Male Age: 20-29
- Cohort 2 (n=10): Gender: Female Age: 20-29
- Cohort 3 (n=10): Gender: Male Age: 30-39
- Cohort 4 (n=10): Gender: Female Age: 30-39
- Cohort 5 (n=10): Gender: Male Age: 40-49
- Cohort 6 (n=10): Gender: Female Age: 40-49
- Cohort 7 (n=10): Gender: Male Age: 50-59
- Cohort 8 (n=10): Gender: Female Age: 50-59

SUMMARY:
Many scientific papers have reported that ERP and QEEG biomarkers can be useful in the evaluation of neurological and psychiatric disorders. A study previously conducted with the COGNISION® system has shown how data collected with the system could help detect cognitive deficits in elderly individuals with probable early Alzheimer's disease (Cecchi et al., 2015). Furthermore, normative ranges for ERP and QEEG parameters are sensitive to subject age (see for example van Dinteren et al., 2014). This study will use advanced EEG techniques to measure brain function among healthy adults ages 20 through 59 to use as reference data to compare against individuals that suffer from neurological and psychiatric disorders. QEEG and ERP parameters from the current study will compliment previously collected normative data in healthy subjects 60 years of age and older (Cecchi et al., 2015).

DETAILED DESCRIPTION:
This is a cross-sectional, observational study in healthy, adult volunteers. This study will use advanced EEG techniques to measure brain function among healthy adults ages 20 through 59 to use as reference data to compare against individuals that suffer from neurological and psychiatric disorders. ERP and QEEG parameters from the current study will complement previously collected normative data in healthy subjects 60 years of age and older (Cecchi et al., 2015).

Study subject population will be stratified by age and gender as detailed in protocol. All assessments will be performed during a single visit that will take up to 90 min. Potential participants will be recruited through local advertising, and participants are free to withdraw from the study at any time. Candidates potentially interested in the study will be explained the purpose of the study, and possible risks and benefits. Those individuals who choose to sign the informed consent will then be screened to ascertain that they meet eligibility. Study subjects that meet inclusion/exclusion criteria will be tested to collect ERP and QEEG parameters using the FDA-cleared COGNISION® system. Data from the ERP and EEG tests will be used to generate ERP and QEEG parameters from the study.

The ERP/EEG testing session will be about 40 min long. Tests administered will include an active, Auditory Oddball ERP test, a Vigilance EEG test, and an Eyes-closed Resting EEG test. A participant may be withdrawn from the study if: 1) The participant fails to meet inclusion/exclusion criteria or 2) The participant or the study Sponsor feels that it is not in the participant's best interest to continue. Upon withdrawal, no further assessments will be performed on the participant and no additional participation will be required of the participant. Additional participants will be recruited to replace withdrawn study subjects, until the study reaches full enrollment of 80 completers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers 20-59 years of age, inclusive.
2. Willingness and ability to provide 1 form of identification with picture.
3. Willingness and ability to provide to understand the requirements of the study, provide written informed consent, and abide by the study procedures.
4. Fluency in English, even if English is not the primary language.
5. Ability to tolerate the electrode cap for the duration of the testing session.
6. Subject has not been enrolled or actively participating in another clinical study 4 weeks prior to testing.

Exclusion Criteria:

1. History of neurological and/or psychiatric disorders:

   * Diseases of the Dementia type (i.e. Alzheimer's Disease, Vascular Dementia, Parkinson's Disease Dementia etc.)
   * Epileptic seizures
   * Bipolar Disorder
   * Autism Spectrum Disorder
   * Depression
   * Brain tumor(s)
   * Multiple Sclerosis
   * Schizophrenia or Schizoaffective Disorder
   * Stroke (ischemic or hemorrhagic)
   * Traumatic Brain Injury
   * Current Drug or Alcohol Abuse
2. Diagnosis with HIV/AIDS
3. Inability to detect a 1000Hz tone at 40dB in either ear.
4. Recent (24 hours) use of medications known to affect QEEG/ERP (cannabinoids, sleep aides, benzodiazepines, opiates/opioids, amphetamines, or barbiturates).
5. Recent (day of study) use of energy drinks, including pre-workout drinks and over the counter energy supplements and nootropics.
6. Caffeine, alcohol, or products containing nicotine within 1 hour of testing.
7. Known allergy to latex.
8. Any impairment, activity, or situation that, in the judgment of the study Sponsor, would prevent satisfactory completion of the study protocol.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Approximately 80 male and female participants between 20 and 59 years of age (inclusive) who meet all eligibility requirements as specified, will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Amplitude for parameters from the Active, Auditory Oddball ERP test. | Day 1
  Amplitude (in microvolts) for the following parameters from the Active, Oddball ERP test:
  1. P50
  2. N100
  3. P200
  4. N200
  5. P3b
Latency for parameters from the Active, Auditory Oddball ERP test. | Day 1
  Latency (in milliseconds) for the following parameters from the Active, Auditory Oddball ERP test:
  1. P50
  2. N100
  3. P200
  4. N200
  5. P3b
Task accuracy from the behavioral response during the Active, Auditory Oddball ERP test. | Day 1
  Change in task accuracy as a percentage of correct behavioral responses during the Active, Auditory Oddball ERP test.
Reaction Time from the behavioral response during the Active, Auditory Oddball ERP test. | Day 1
  Median reaction time for the correct behavioral responses measured in milliseconds during the Active, Auditory Oddball ERP test.
QEEG measures from the Vigilance EEG | Day 1
  Changes in Absolute Power (measured in µv2/Hz) for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
  * Gamma power
  * Total power
QEEG measures from the Eyes-closed Resting EEG | Day 1
  Changes in Absolute Power (measured in µv2/Hz) for the following Pharmaco-EEG parameters:
  * Delta power
  * Theta power
  * Alpha power
  * Beta power
  * Gamma power
  * Total power
  * Changes in frequency (measured in Hz) for peak alpha

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cecchi, PhD, Principal Investigator — COGNISION
Locations (1):
- Cognision, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cecchi M, Adachi M, Basile A, Buhl DL, Chadchankar H, Christensen S, Christian E, Doherty J, Fadem KC, Farley B, Forman MS, Honda S, Johannesen J, Kinon BJ, Klamer D, Marino MJ, Missling C, O'Donnell P, Piser T, Puryear CB, Quirk MC, Rotte M, Sanchez C, Smith DG, Uslaner JM, Javitt DC, Keefe RSE, Mathalon D, Potter WZ, Walling DP, Ereshefsky L. Validation of a suite of ERP and QEEG biomarkers in a pre-competitive, industry-led study in subjects with schizophrenia and healthy volunteers. Schizophr Res. 2023 Apr;254:178-189. doi: 10.1016/j.schres.2023.02.018. Epub 2023 Mar 13. PMID 36921403
- [Result] Cecchi M, Moore DK, Sadowsky CH, Solomon PR, Doraiswamy PM, Smith CD, Jicha GA, Budson AE, Arnold SE, Fadem KC. A clinical trial to validate event-related potential markers of Alzheimer's disease in outpatient settings. Alzheimers Dement (Amst). 2015 Oct 2;1(4):387-94. doi: 10.1016/j.dadm.2015.08.004. eCollection 2015 Dec. PMID 27239520
- [Result] Haller, M., Donoghue, T., Peterson, E., Varma, P., Sebastian, P., Gao, R., … Voytek, B. (2018). Parameterizing neural power spectra. BioRxiv, 299859. https://doi.org/10.1101/299859
- [Result] Jobert M, Wilson FJ, Ruigt GS, Brunovsky M, Prichep LS, Drinkenburg WH; IPEG Pharmaco-EEG Guidelines Committee. Guidelines for the recording and evaluation of pharmaco-EEG data in man: the International Pharmaco-EEG Society (IPEG). Neuropsychobiology. 2012;66(4):201-20. doi: 10.1159/000343478. Epub 2012 Oct 12. PMID 23075830
- [Result] van Dinteren R, Arns M, Jongsma ML, Kessels RP. P300 development across the lifespan: a systematic review and meta-analysis. PLoS One. 2014 Feb 13;9(2):e87347. doi: 10.1371/journal.pone.0087347. eCollection 2014. PMID 24551055